CLINICAL TRIAL: NCT01965769
Title: Effects Of Not Measuring Gastric Residuals Prior To Enteral Bolus Feeding On Gastrointestinal Function And Feeding Tolerance In Very Low Birth Weight Infants
Brief Title: Effects Of Not Measuring Gastric Residual Content On Feeding Tolerance In Premature Infants iNFANTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-216; Gerber003 (Other: Gerber)
Record Dates: First submitted 2013-10-15; First posted 2013-10-18 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-10

CONDITIONS: Premature Infant
Keywords: Very low birth weight infants; premature; nutrition; gastric residual
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- no gastric residual evaluation (Experimental): Infants will not receive routine gastric residual evaluation prior to feeding
  Interventions: Other: No gastric residual evaluation
- gastric residual evaluation (No Intervention): Infants will receive routine gastric residual evaluation

INTERVENTIONS:
Other: No gastric residual evaluation — Infants will not receive routine gastric residual evaluation prior to feeding.
  Arms: no gastric residual evaluation

SUMMARY:
Omitting evaluation of gastric residual contents prior to feeding very premature infants will increase the feeding intake at 2 weeks, and total caloric intake and growth by 3 weeks, as well as decrease the time required for parenteral nutrition.

DETAILED DESCRIPTION:
Infants were randomized into 2 groups. Group 1 had no gastric residuals evaluated prior to feeding. Group 2 had gastric residuals evaluated prior to feeding. Nutritional outcomes were compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age less than 32 weeks,
* Birth weight less than or equal to 1250 grams,
* Initial feeding tolerated within 48 hours of life

Exclusion Criteria:

* Congenital or chromosomal disorders,
* Severe complications leading to death in the first week of life

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2011-03; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Amount of feeding intake at 2 weeks | Baseline to 2 weeks

SECONDARY OUTCOMES:
Days to 120 mL/kg/d of enteral feedings | Baseline to approximately 21 days
Days of parenteral nutrition | Baseline to approximately 21 days
Incidence of late onset sepsis | Baseline to approximately 90 days
Weekly or biweekly liver function tests | Baseline to 42 days
  Direct bilirubin
Growth indices | Baseline to approximately 90 days
  Weight, length and head circumference
Length of hospital stay | Baseline to approximately 90 days
Incidence of necrotizing enterocolitis | Baseline to approximately 90 days
Days requiring a central venous line | Baseline to approximately 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Josef Neu, MD, Principal Investigator — University of Florida
Locations (1):
- UF & Shands Hospital, Gainesville, Florida, United States